CLINICAL TRIAL: NCT02923232
Title: Ocular Adaptation and Visual Performance for Accommodative Contact Lens
Acronym: ACL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding organization requested to stop the study
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Shun-nan Yang, Director of Research at VPI, Pacific University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OFV-S1
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Functionality of Experimental Contact Lens
Keywords: Contact lens; Accommodation; Visual performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accommodative contact lens (Experimental): The accommodative contact lens is composed of traditional hydrogel lens material but has an internal cavity to allow lens deformation that increases its refractive power at an downward angle.
  Interventions: Device: Accommodative contact lens

INTERVENTIONS:
Device: Accommodative contact lens — Different downgaze angles will be experimented to determine whether the accommodative contact lens can alter its optical refraction at downgaze angles.

SUMMARY:
Presbyopes (people who might have a significant loss of their ability to accommodate their crystalline lens in the eye) will be recruited to wear a test lens and perform typical clinical tests of visual acuity with different luminance levels and viewing distances/angles.

DETAILED DESCRIPTION:
In the proposed study we plan to recruit presbyopes (people who might have a significant loss of their ability to accommodate their crystalline lens in the eye) to wear a test lens and perform typical clinical tests of visual acuity with different luminance levels and viewing distances/angles. These are similar to the typical examinations conducted for regular contact lens wearers. Results of this testing will be used to evaluate the efficacy of test lenses and to provide additional information for revision of test lenses. If shown to provide adequate eye comfort and intended vision correction, this lens design has the potential of allowing tens of millions of presbyopes to adapt to contact lenses and significantly improve their vision and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Be between 40 and 65 years of age.
* Have normal/corrected-to-normal monocular acuity of better than 20/25 for both eyes.
* Have pupil diameter in regular lighting ≥ 2.5 mm.
* Willing and able to wear multifocal contact lenses in both eyes.
* Have a current optical prescription (obtained less than 2 years ago).
* Have spherical equivalent correction equal to or higher than -1.00 Diopter and equal to or less than +0.50 Diopter.
* Have cylindrical correction equal to less than 0.50 Diopter.

Exclusion Criteria:

* Have no prismatic correction.
* Without any eye infection, inflammation, disease, or abnormality that contraindicates contact lens wear within the past 6 months.
* No clinically significant ocular pathology (e.g., cataract, keratoconus, dry eye, diabetic retinopathy, or age-related macular degeneration)
* Have no photosensitive disorders, including migraine and seizure.
* Have no binocular dysfunction, including amblyopia, strabismus, and other binocular diseases.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-11; Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Performance Institute, Forest Grove, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study involved few participants recruited from Pacific University and designated clinics. It went through 3 iterations in lens design changes and less than 10 subjects in each iteration.
Pre-assignment Details: Subjects were recruited in 3 separate iterations. They were not assigned to different groups, and were tested with the same test lens with minor modification. This is considered a phase 1 study.
Groups:
- Accommodative Contact Lens: This was a study involving only the test contact lens. There is no control condition.
Period: Overall Study
Arm/Group | Accommodative Contact Lens
Started | 52
Completed | 52 (The study was not completed due to the withdraw of research funding.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Presbyopes
Units Other Than Participants: eyes
Arm/Group | Accommodative Contact Lens
Number analyzed (Participants) | 52
Number analyzed (eyes) | 52
Age, Customized [Mean (Standard Deviation); unit: year]
  Age at the entrance date | 52.6 (14.2)
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 32
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Monocular visual acuity [Mean (Standard Deviation); unit: logMAR] — Subjects wore no optical correction and their distance monocular acuity was assessed.
  logMAR | .4 (.23)

OUTCOME MEASURES:

1. Primary Outcome: Monocular Refractive Power
Description: Participants will wear the test lens and look at different downsize angles. The refractive power of the lens/eye combination will be measured with an open-field auto refractor.
Time Frame: 30 mins of wearing; non-dispensing.
Population: Presbyopes who require distance optical correction
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: eyes
Arm/Group | Accommodative Contact Lens
Number analyzed (Participants) | 52
Number analyzed (eyes) | 52
Diopter | -1.5 (2.42)

2. Primary Outcome: Visual Acuity at 20 Degree Downsize Angles
Description: The resultant visual acuity at near at this down-gaze angle will be measured. This is achieved by having the subjects holding a new acuity chart at 40 cm distance, their heads upright and perpendicular to the ground, and their gazes rotated downward 20 degrees where the chart was located. The subjects then read out the optotypes (letters) on the chart to a size they cannot no only identify the letters. The lines of letters with which all letters can be identified is recorded as the corresponding level of acuity.
Time Frame: 30 mins of wearing; non-dispensing.
Population: Presbyopes who require distance optical correction
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Accommodative Contact Lens
Number analyzed (Participants) | 52
logMAR | 0.24 (0.22)

ADVERSE EVENTS:
Time Frame: Duration of wear, usually no more than 30 mins.
Description: This is a non-prescription study involving only temporarily worn contact lens for a period of 30 mins during which refractive error and acuity of tested eyes were measured. As such, there is no expected risk in mortality and serious adverse effects.
Arm/Group | Accommodative Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02923232/Prot_ICF_000.pdf